CLINICAL TRIAL: NCT03191318
Title: Randomized Control Trial to Compare the Outcomes of Enhanced Recovery After Surgery (ERAS) Pathway and Standard Recovery Pathway After Laparoscopic Sleeve Gastrectomy
Brief Title: Comparison of Enhanced Recovery After Surgery (ERAS) Pathway With Conventional Pathway After Laparoscopic Sleeve Gastrectomy
Acronym: BARI-ERAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GEM Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BARI-01
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Morbid Obesity
Keywords: ERAS; Enhanced recovery after sugery in bariatric surgery; sleeve gastrectomy
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS pathway (Active Comparator): Laparoscopic sleeve gastrectomy with ERAS pathway
  Interventions: Other: ERAS pathway
- Standard pathway (Active Comparator): Laparoscopic sleeve gastrectomy with standard pathway
  Interventions: Other: Standard pathway

INTERVENTIONS:
Other: ERAS pathway — ERAS pathway after laparoscopic sleeve gastrectomy
  Other Names: Fast track pathway
  Arms: ERAS pathway
Other: Standard pathway — Standard pathway after laparoscopic sleeve gastrectomy
  Other Names: Coventional pathway
  Arms: Standard pathway

SUMMARY:
The aim of this study is to compare two postoperative recovery pathways namely, enhanced recovery after surgery (ERAS) pathway and conventional recovery pathway after laparoscopic sleeve gastrectomy with respect to outcomes including hospital stay, postoperative pain and other postoperative outcomes.

DETAILED DESCRIPTION:
The Enhanced recovery after surgery (ERAS) pathway, initially introduced for colorectal surgery, is an evidence based perioperative pathway which has resulted in earlier recovery, less pain, and lower complication rates. Bariatric surgical patients, without severe co-morbidities, are good candidates for ERAS pathway, but the application of ERAS concepts has been limited in this field, specially, in Asia.

Although the current literature shows that 2 randomized clinical trials (RCT) have been performed for application of ERAS in bariatric surgery, data is still scarce as per outcomes with respect to postoperative pain and analgesic usage. One of the RCTs has compared with historical controls and both the RCTs have not clearly defined their conventional standard pathways. In this study, the investigators have clearly defined both ERAS pathway and standard pathway leaving no ambiguity.

This study is a prospective, randomized, parallel group trial comparing ERAS pathway and standard pathway after laparoscopic sleeve gastrectomy in relation to the hospital stay, postoperative pain, complications and other perioperative parameters.

This is a single institute based trial, being conducted at GEM hospital and research centre, Coimbatore, TN, India. The trial has been approved by the GEM Hospital ethical committee.

In this trial, the investigators are planning to enroll participants with morbid obesity planned to undergo laparoscopic sleeve gastrectomy. After full assessment, informed consent, these participants will be randomised using computer generated random numbers either into ERAS pathway group or into Standard pathway group.

All the intraoperative and perioperative details with respect to anaesthetic drugs usage, intravenous fluid requirement, time to ambulation, time to oral liquids, postoperative pain score, analgesic requirement and hospital stay will be recorded in the proforma.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing laparoscopic sleeve gastrectomy during this study period

Exclusion Criteria:

* 1. Redo procedures 2. ASA III and above status 3. Previous major upper abdominal surgeries 4. Not willing to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Hospital stay | 7 days
  Postoperative hospital stay of patients

SECONDARY OUTCOMES:
Pain score | Within 72 hours of surgery
  Postoperative pain score
Operative time | Within 24 hours, in minutes
  Time taken to perform surgery
Analgesic requirement | Within 72 hours
  Post operative cumulative analgesic requirement
Complication rate | Within 30 days
  Post operative complications rate

CONTACTS AND LOCATIONS:
Overall Officials: C Palanivelu, MS, MCh, Study Chair — GEM Hospital & Research centre; P Praveen Raj, MS, DNB, Study Director — GEM Hospital and Research centre; M S Prabhakaran, DA, Principal Investigator — GEM Hospital & Research centre; Siddhartha Bhattacharya, MS, DNB, FNB, Principal Investigator — GEM Hospital & Research centre
Locations (1):
- Gem Hospital and Research Centre, Coimbatore, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No
It may be obtained by request

REFERENCES:
- [Background] Pimenta GP, Capellan DA, de Aguilar-Nascimento JE. Sleeve Gastrectomy With or Without a Multimodal Perioperative Care. A Randomized Pilot Study. Obes Surg. 2015 Sep;25(9):1639-46. doi: 10.1007/s11695-015-1573-2. PMID 25670530
- [Background] Lemanu DP, Singh PP, Berridge K, Burr M, Birch C, Babor R, MacCormick AD, Arroll B, Hill AG. Randomized clinical trial of enhanced recovery versus standard care after laparoscopic sleeve gastrectomy. Br J Surg. 2013 Mar;100(4):482-9. doi: 10.1002/bjs.9026. Epub 2013 Jan 21. PMID 23339040
- [Derived] Prabhakaran S, Misra S, Magila M, Kumar SS, Kasthuri S, Palanivelu C, Raj PP. Randomized Controlled Trial Comparing the Outcomes of Enhanced Recovery After Surgery and Standard Recovery Pathways in Laparoscopic Sleeve Gastrectomy. Obes Surg. 2020 Sep;30(9):3273-3279. doi: 10.1007/s11695-020-04585-2. PMID 32291702